CLINICAL TRIAL: NCT01893086
Title: Impact of Opportunistic Salpingectomy on Ovarian Reserve in Patients Undergoing Laparoscopic Hysterectomy: a Multi-center, Randomized Controlled Trial
Brief Title: Impact of Opportunistic Salpingectomy on Ovarian Reserve in Patients Undergoing Laparoscopic Hysterectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CHA University (Other)
Responsible Party: Principal Investigator, Taejong Song, Professor, CHA University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KNC13-029
Record Dates: First submitted 2013-07-02; First posted 2013-07-08 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Benign Uterine Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LH alone (Active Comparator): LH, laparoscopic hysterectomy
  Interventions: Procedure: LH alone
- LH with opportunistic salpingectomy (Experimental): LH, laparoscopic hysterectomy
  Interventions: Procedure: LH with opportunistic salpingectomy

INTERVENTIONS:
Procedure: LH alone — LH, laparoscopic hysterectomy
  Arms: LH alone
Procedure: LH with opportunistic salpingectomy — LH, laparoscopic hysterectomy
  Arms: LH with opportunistic salpingectomy

SUMMARY:
Recently, many gynecologic oncologists proposed that surgeons should consider opportunistic salpingectomy to prevent ovarian cancer for all patients undergoing hysterectomy for benign disease. However, the safety and the consequences regarding ovarian function after salpingectomy have not yet to be established. Therefore, the aim of this randomized controlled study is compare the ovarian reserve via anti-Müllerian hormone (AMH) between laparoscopic hysterectomy (LH) alone and LH combined with salpingectomy.

ELIGIBILITY:
Inclusion Criteria:

* women who were planning to undergo laparoscopic hysterectomy for benign uterine diseases
* women aged between 19 and 52 years
* women with regular menstruation (defined as the duration of menstrual cycle between 21 and 45 days)
* women who were appropriated medical status for laparoscopic surgery

Exclusion Criteria:

* any ovarian cysts requiring ovarian surgery
* any suspicious findings of malignant diseases
* history of prior salpingectomy or salpingo-oophorectomy
* pregnant or menopausal status
* preoperative serum anti-Müllerian hormone (AMH) < 0.30 ng/mL
* use of hormonal treatments in the three months before surgery
* any other endocrine disease (such as uncontrolled thyroid dysfunction, hyperprolactinemia, or Cushing syndrome)
* an inability to understand and provide written informed consent.

Ages: 19 Years to 52 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2013-06; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change in ovarian reserve | 3 months after surgery
  The primary outcome measure was the change of ovarian reserve, determined by the rate of decline in AMH level from before surgery to 3-month post-surgery with the following formula : decline rate (%) = 100 × (preoperative AMH level - postoperative AMH level) ÷ preoperative AMH level.

CONTACTS AND LOCATIONS:
Overall Officials: Taejong Song, MD PhD, Principal Investigator — Kangbuk Samsung Hospital, Seoul, Republic of Korea
Locations (3):
- South Korea (3):
  - Keimyung University School of Medicine, Daegu
  - Kangbuk Samsung Hospital, Seoul
  - CHA Gangnam Medical Center, Seoul